CLINICAL TRIAL: NCT00915850
Title: Phase I/II Trial of Combination Chemotherapy With Docetaxel, Cisplatin and 5-FU for Unresectable Advanced Esophageal Cancer.
Brief Title: Trial of Docetaxel, Cisplatin, Fluorouracil (5-FU) for Unresectable Advanced Esophageal Squamous Cell Carcinoma (ESCC)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wakayama Medical University (Other)
Responsible Party: Makoto Iwahasi, Wakayama Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WMU-EC01
Record Dates: First submitted 2009-06-05; First posted 2009-06-08 (Estimated); Last update posted 2010-09-09 (Estimated); Status verified 2010-09

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Anticancer drug (Experimental): docetaxel, cisplatin and 5-FU
  Interventions: Drug: DCF

INTERVENTIONS:
Drug: DCF — docetaxel, Cisplatin and 5-FU
  Other Names: docetaxel+Cisplatin+5-FU

SUMMARY:
This phase I/II study is being conducted to determine the maximum-tolerated dose (MTD), dose-limiting toxicity (DLT), and efficacy of a combination chemotherapy using docetaxel, cisplatin and 5-fluorouracil (DCF) in unresectable advanced esophageal cancer. The usefulness of the this regimen is evaluated by RECIST, time to progression and median survival time.

DETAILED DESCRIPTION:
<Phase I>

Primary Objective:

To establish the safety of combination chemotherapy comprising docetaxel (escalating doses: 25,30,35,40 mg/m2,day1 and day8), cisplatin (12mg/m2,day1-5), and fluorouracil (600mg/m2,day1-5) (DCF) in unresectable advanced esophageal cancer.

Secondary Objective:

To observe the efficacy of this regimen in these patients.

<Phase II>

Primary Objective:

To assess the response rate of combination chemotherapy comprising docetaxel (recommended dose determined in phase I study,day1 and day8), cisplatin (12 mg/m2, day1-5), and fluorouracil (600 mg/m2, day1-5) (DCF) in unresectable advanced esophageal cancer.

Secondary Objectives:

To determine the adverse reactions of this regimen in these patients. To determine TTP(Time to progression) of patients treated with this regimen. To determine MST(Median survival time) of patients treated with this regimen.

ELIGIBILITY:
Inclusion Criteria:

* locally advanced or metastatic esophageal cancer precluding curative surgical resection and recurrent esophageal cancer measurable disease by CT scan
* ECOG performance status 0-1
* 20 years and older
* Patients must have clinically documented unresectable or metastatic esophageal cancer and histologic confirmation of the diagnosis with tumor
* Tissue from tumor must be available
* Patients must have measurable disease
* Patients may have received prior adjuvant chemotherapy; this must have been completed at least 1 month
* Life expectancy > 3 months
* Laboratory values as follows
* 3000/mm3 < WBC < 12000/mm3
* 1500/mm3 < granulocyte count
* 8.0 gm/dl < hemoglobin
* Platelet count > 100000/mm3
* Aspartate transaminase < 150 IU/L
* Alanine transaminase < 150 IU/L
* Creatinine < 1.5 mg/dl
* Able and willing to give valid written informed consent

Exclusion Criteria:

* Pregnancy (women of childbearing potential: refusal or inability to use effective means of contraception)
* Active or uncontrolled infection
* Prior chemotherapy or radiation therapy within 4 weeks, surgery within 3 weeks or immunotherapy within 1 week
* Clinically significant heart disease
* Patients with a history of myocardial infarction within the previous three months
* Patients with uncontrolled diabetes mellitus or hypertension
* Presence of clinically apparent central nervous system metastases
* Patients with any other severe concurrent disease, which in the judgment of the investigator, would make the patient inappropriate for entry into this study
* Decision of unsuitableness by principal investigator or physician-in-charge

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2007-08; Primary Completion 2010-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Safety (Phase I: toxicities as assessed by NCI CTCAE version3) and efficacy (Phase II: Feasibility as evaluated by RECIST) | 1 month

SECONDARY OUTCOMES:
To determine the recommended phase II dose of docetaxel (Phase I) | 1 month
To determine the clinical effectiveness in the patients with measurable disease (Phase I) | 1 month
To analyze the toxicity (Phase II) | 1 month
Time to progression (Phase II) | 5 years
median survival time (Phase II) | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Makoto Iwahashi, M.D., Study Director — Second Department of Surgery, Wakayama Medical University
Locations (1):
- Wakayama Medical University, Wakayama, Wakayama, Japan